CLINICAL TRIAL: NCT02400918
Title: Self-help for Treating Social Anxiety Disorder: An Evaluation of a Mindfulness and Acceptance-based Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Meagan MacKenzie, Postdoctoral Fellow, Wilfrid Laurier University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WilfridLU
Record Dates: First submitted 2015-03-23; First posted 2015-03-27 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Anxiety; Shyness
MeSH Terms: conditions — Anxiety Disorders; Shyness

ARMS (2):
- Workbook (Experimental): They will be directed to use the 8-week plan included in The Mindfulness and Acceptance-based Workbook for Social Anxiety and Shyness (Fleming & Kocovski, 2013), an ACT-based self-help book and to access mindfulness audio files located on the publisher's website (as described in the book).
  Interventions: Other: The Mindfulness and Acceptance-based Workbook for Social Anxiety and Shyness (Fleming & Kocovski, 2013)
- Control (No Intervention): Waitlist control

INTERVENTIONS:
Other: The Mindfulness and Acceptance-based Workbook for Social Anxiety and Shyness (Fleming & Kocovski, 2013) — An acceptance and commitment therapy-based self-help workbook for social anxiety and shyness. It includes an 8-week program.
  Arms: Workbook

SUMMARY:
Social anxiety disorder (SAD) is the most common anxiety disorder, affecting up to 10% of the population and causing significant distress. Fortunately, there are effective interventions including cognitive behavior therapy (CBT) and acceptance and commitment therapy (ACT). However, only about a third of people with SAD seek treatment. There are a number of barriers to seeking treatment, including cost, availability, and stigma. Self-help may be one way to reach people who may not otherwise present for treatment. Research on self-help books for SAD based on CBT has yielded promising results. However, no research to date has examined the efficacy of ACT-based self-help for SAD. The primary purpose of the present study is to evaluate The Mindfulness and Acceptance-based Workbook for Social Anxiety and Shyness (Fleming & Kocovski, 2013), an ACT-based self-help book. Socially anxious participants will be randomly assigned to receive the workbook or be placed on a waitlist. It is hypothesized that workbook participants will report significantly reduced social anxiety at the end of eight weeks compared to waitlist participants. The secondary purpose is to evaluate how the treatment works. Increases in mindfulness and acceptance have been shown to lead to reduced social anxiety. These same variables will be examined in the present study. Finally, this research aims to examine variables that can predict who may do well in treatment. Given that two-thirds of people who meet criteria for this disorder will not seek traditional treatments, it is important to develop and evaluate alternative treatments, including those based on self-help.

ELIGIBILITY:
Inclusion Criteria:

* must be seeking help for shyness/social anxiety

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 4 and 8 weeks later in The Liebowitz Social Anxiety Scale (Liebowitz, 1987) | Baseline and 4 weeks and 8 weeks
  Self-reported social anxiety scores. Each item is scored 0 (none) to 3 (severe) yielding a total between 0 and 72.
Change from Baseline to 4 and 8 weeks later in the Freiberg Mindfulness Inventory (Buchheld, Grossman, & Walach, 2001) | Baseline and 4 weeks and 8 weeks
  Self-reported mindfulness. Each item is scored 0 (rarely) to 4 (almost always) yielding a total between and 0 and 56.
Change from Baseline to 4 and 8 weeks later in the Social Anxiety - Acceptance and Action Questionnaire (MacKenzie & Kocovski, 2010) | Baseline and 4 weeks and 8 weeks
  Self-reported acceptance of social anxiety symptoms. Each item is scored 1 (never true) to 7 (always true) yielding a total between and 19 and 133.
Change from Baseline to 4 and 8 weeks later in the Beck Depression Inventory (Beck, Steer, & Brown, 1996) | Baseline and 4 weeks and 8 weeks
  Self-reported depression symptoms. Each item is scored 0 to 3 yielding a total between and 0 and 63.
Treatment credibility will be assessed using the scale by Devilly and Borkovec (2000) one week following the start of treatment (consistent with Nordgreen et al., 2012). | One week following the start of treatment
  This 6-item scale assesses the participants' idea of treatment credibility.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Kocovski, PhD, Principal Investigator — Wilfrid Laurier University
Locations (1):
- Wilfrid Laurier University, Waterloo, Ontario, Canada